CLINICAL TRIAL: NCT02973100
Title: A Phase 2, Double-Blind, Placebo-Controlled, 18-Week Trial of Investigational Dulaglutide Doses Versus Placebo in Patients With Type 2 Diabetes on Metformin Monotherapy
Brief Title: A Study of Investigational Dulaglutide Doses in Participants With Type 2 Diabetes on Metformin Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16568; H9X-MC-GBGJ (Other: Eli Lilly and Company); 2016-002494-34 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Dulaglutide 4.5mg (Experimental): 4.5mg of Dulaglutide administered subcutaneously (SC)
  Interventions: Drug: Dulaglutide
- Dulaglutide 3.0mg (Experimental): 3.0mg of Dulaglutide administered SC
  Interventions: Drug: Dulaglutide
- Dulaglutide 1.5mg (Active Comparator): 1.5mg of Dulaglutide administered SC
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: Dulaglutide 1.5mg; Dulaglutide 3.0mg; Dulaglutide 4.5mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of investigational doses of dulaglutide in participants with type 2 diabetes on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have had type 2 diabetes (T2D) for ≥6 months according to the World Health Organization (WHO) classification
* Have HbA1c of 7.0% to 10.0%, inclusive, as assessed by the central laboratory
* Have been treated with stable doses of metformin for at least 3 months
* Have a body mass index (BMI) ≥25 kilograms per square meter

Exclusion Criteria:

* Have type 1 diabetes (T1D)
* Have used any glucose-lowering medication other than metformin 3 months prior to study entry or during screening/lead-in period or have used any glucagon-like peptide-1 receptor agonists (GLP-1 RAs) at any time in the past
* Have had any of the following cardiovascular conditions: acute myocardial infarction (MI), New York Heart Association Class III or Class IV heart failure, or cerebrovascular accident (stroke)
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial
* Have had chronic or acute pancreatitis any time prior to study entry
* Have an estimated glomerular filtration rate (eGFR) <45 milliliters/minute/1.73 square meter, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation
* Have serum calcitonin ≥20 picograms per milliliter, as determined by the central laboratory at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07-15 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (38):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - Marin Endocrine Associates, Greenbrae, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley Lake, California
  - University Clinical Investigators, Inc., Tustin, California
  - Infosphere, Van Nuys, California
  - Diablo Clinical Research, Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Axes Medical Research, LLC, Cooper City, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Research Group, LLC, Miami Lakes, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - In-Quest Medical Research, LLC - Norcross, Norcross, Georgia
  - East West Medical Institute, Honolulu, Hawaii
  - Elite Cilnical Trials LLLP, Blackfoot, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - HSHS Medical Group Diabetes Research, Springfield, Illinois
  - American Health Network, Indianapolis, Indiana
  - Iderc, P.L.C., Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Manhattan Medical Research, New York Mills, New York
  - High Point Clinical Trials Center, High Point, North Carolina
  - Aventiv Research, Columbus, Ohio
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - New Phase Research & Development, Knoxville, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Consano Clinical Research, San Antonio, Texas
  - Clinpoint Trial, LLC, Waxahachie, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Rainier Clinical Research Center, Renton, Washington
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandýs nad Labem-Stará Boleslav
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Praha 4 - Krc
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ruda Śląska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- Puerto Rico (2):
  - Marginal Doctor's Center, Manatí
  - American Telemedicine Center, San Juan
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alba Iulia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Satu Mare

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Investigational Dulaglutide Doses in Participants With Type 2 Diabetes on Metformin Monotherapy — https://www.lillytrialguide.com/en-US/studies/type-2-diabetes/GBGJ#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 3 periods: an approximately 2-week lead-in period, followed by an 18-week treatment period, and a 4-week safety follow-up period.
Groups:
- Placebo: Participants received placebo once weekly (QW) by subcutaneous (SC) injection.
- Dulaglutide 1.5 Milligrams (mg): Participants received 1.5mg of dulaglutide QW by SC injection.
- Dulaglutide 3.0mg: Participants received 3.0mg of dulaglutide QW by SC injection.
- Dulaglutide 4.5mg: Participants received 4.5mg of dulaglutide QW by SC injection.
Period: Overall Study
Arm/Group | Placebo | Dulaglutide 1.5 Milligrams (mg) | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Started | 82 | 81 | 79 | 76
Received at Least 1 Dose of Study Drug | 81 | 81 | 79 | 76
Completed | 75 | 73 | 75 | 69
Not Completed | 7 | 8 | 4 | 7
Not completed — Adverse Event | 1 | 2 | 1 | 2
Not completed — Lost to Follow-up | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 1 | 4
Not completed — Notification of change in address | 0 | 0 | 0 | 1
Not completed — Failed to attend Safety followup period | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dulaglutide 1.5mg: Participants received 1.5mg of dulaglutide QW by SC injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg | Total
Number analyzed (Participants) | 81 | 81 | 79 | 76 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.52 (8.93) | 57.65 (9.79) | 55.90 (10.74) | 57.13 (9.63) | 56.80 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 44 | 40 | 159
  Male | 48 | 39 | 35 | 36 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 32 | 38 | 30 | 135
  Not Hispanic or Latino | 46 | 49 | 40 | 45 | 180
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 6 | 9 | 6 | 31
  Asian | 0 | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 6 | 6 | 6 | 6 | 24
  White | 59 | 68 | 58 | 59 | 244
  More than one race | 5 | 1 | 4 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 6 | 6 | 5 | 4 | 21
  United States | 42 | 45 | 44 | 43 | 174
  Czechia | 10 | 9 | 10 | 8 | 37
  Poland | 13 | 11 | 10 | 10 | 44
  Mexico | 10 | 10 | 10 | 11 | 41
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of glycosylated hemoglobin | 8.08 (0.79) | 8.02 (0.80) | 8.16 (0.92) | 8.12 (0.81) | 8.09 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with baseline as a covariate, pooled country, treatment, time, treatment*time as fixed effects.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had postbaseline values, excluding post rescue data for Hemoglobin A1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 70 | 73 | 73 | 66
Percentage of glycosylated hemoglobin | -0.44 (0.101) | -1.23 (0.099) | -1.31 (0.099) | -1.40 (0.103)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide 1.5mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.07 to -0.53]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide 3.0mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.14 to -0.60]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide 4.5mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.24 to -0.69]

2. Secondary Outcome: Percentage of Participants With HbA1c of <7.0%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 18
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 70 | 73 | 73 | 66
Percentage of Participants | 20 | 71.2 | 71.2 | 68.2
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide 1.5mg; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 24.489, 95% CI 2-sided [8.368 to 71.667]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide 3.0mg; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 27.906, 95% CI 2-sided [9.238 to 84.300]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide 4.5mg; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 21.852, 95% CI 2-sided [7.672 to 62.242]

3. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: Fasting serum glucose (FSG) is a test to determine how much glucose (sugar) is in a serum sample after an overnight fast. Least Squares (LS) means was determined by MMRM methodology with baseline as a covariate, pooled country, baseline HbA1c strata using >=8% as cutoff, treatment, time, treatment*time as fixed effects.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had postbaseline values, excluding post rescue data for FSG.
Measure: Least Squares Mean (Standard Error); unit: millimole/liter (mmol/L)
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 63 | 62 | 67 | 61
millimole/liter (mmol/L) | -0.69 (0.257) | -2.01 (0.261) | -1.92 (0.250) | -2.11 (0.263)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide 1.5mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-2.02 to -0.62]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide 3.0mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.91 to -0.54]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide 4.5mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-2.12 to -0.72]

4. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with baseline as a covariate, pooled country, baseline HbA1c strata using >=8% as cutoff, treatment, time, treatment*time as fixed effects.
Time Frame: Baseline, Week 18
Population: All randomized participants who received at least one dose of study drug and had postbaseline values, excluding post rescue data for body weight.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (Kg)
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 70 | 72 | 74 | 67
Kilograms (Kg) | -1.6 (0.39) | -2.8 (0.39) | -3.9 (0.39) | -4.1 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Dulaglutide 1.5mg; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs Dulaglutide 3.0mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.4 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs Dulaglutide 4.5mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-3.7 to -1.5]

5. Secondary Outcome: Percentage of Participants Discontinuing Study Drug Due to Adverse Events
Description: Adverse event (AE) defined as any unfavorable medical event, newly emerged or a deterioration of a preexisting condition, in other words any untoward medical occurrence in a patient administered a pharmaceutical product, without regard to the possibility of a causal relationship, that occurred after the visit for informed consent and up to the visit for completion of administration, or discontinuation.
Time Frame: Baseline through Week 18
Population: All randomized participants who received study drug and had postbaseline data for safety analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 82 | 81 | 79 | 76
Percentage of Participants | 4.9 | 6.2 | 10.1 | 13.2

6. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemia
Description: Hypoglycemic events (HE) were classified as severe, documented symptomatic (defined as an HE with typical symptoms of hypoglycemia and a blood glucose level of ≤3.9 millimoles per liter [mmol/L]). Hypoglycemia rate per 30 days was summarized at each visit by treatment group. The rate of hypoglycemia was analyzed using a generalized estimation equations model with a negative binomial distribution and a Log link. LS mean was determined by MMRM methodology with baseline hypoglycemia rate, pooled country, HbA1c at Baseline, treatment, with log of exposure in days divided by 365.25 as the offset.
Time Frame: Week 18
Population: All randomized participants who received at least one dose of study drug and had postbaseline values, excluding post rescue values for hypoglycemic episodes.
Measure: Least Squares Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 81 | 81 | 79 | 76
Episodes/participant/365.25 days | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.001)

7. Secondary Outcome: Pharmacokinetics (PK): The Maximum Drug Concentration at Steady State (Cmax,ss) of Dulaglutide
Description: Plasma samples for PK analysis were combined measure obtained from 0, 2, 4, 6, 10, 18, 22 weeks and until early termination of the visit. Cmax takes all time points post dose into account and one value was reported.
Time Frame: 0, 2, 4, 6, 10, 18, 22 weeks and early termination
Population: All randomized participants who received at least one dose of the study drug and have evaluable PK data.
Measure: Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 81 | 79 | 76
nanogram per milliliter (ng/mL) | 90.4 [38.9 to 170] | 151 [64.3 to 277] | 204 [87.2 to 377]

8. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve at Steady State From Time Zero to 168 Hours (AUC[0-168], ss) of Dulaglutide
Description: AUC[0-168h] is a combined measure obtained from 0, 2, 4, 6, 10, 18, 22 weeks and until early termination of the visit.
Time Frame: 0, 2, 4, 6, 10, 18, 22 weeks and early termination
Population: All randomized participants who received at least one dose of the study drug and have evaluable PK data.
Measure: Mean (90% Confidence Interval); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
Number analyzed (Participants) | 81 | 79 | 76
nanogram*hour per milliliter (ng*h/mL) | 11800 [5300 to 21300] | 26700 [15300 to 41400] | 36600 [21100 to 56500]

ADVERSE EVENTS:
Time Frame: Up to 22 weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Placebo | Dulaglutide 1.5mg | Dulaglutide 3.0mg | Dulaglutide 4.5mg
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 0/79 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/81 | 3/81 | 7/79 | 3/76
Other Adverse Events (participants affected / at risk) | 29/81 | 36/81 | 49/79 | 39/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Dulaglutide 1.5mg (N=81) | Dulaglutide 3.0mg (N=79) | Dulaglutide 4.5mg (N=76)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Dulaglutide 1.5mg (N=81) | Dulaglutide 3.0mg (N=79) | Dulaglutide 4.5mg (N=76)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 7 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 9 (17) | 18 (34) | 16 (32)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (10) | 5 (5) | 8 (13)
Eructation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 18 (45) | 20 (32) | 23 (40)
Vomiting (Gastrointestinal disorders) | 4 (6) | 9 (20) | 9 (15) | 10 (16)
Fatigue (General disorders) | 2 (3) | 1 (1) | 4 (4) | 7 (7)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (1) | 5 (5) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 5 (7) | 2 (2) | 6 (6) | 3 (4)
Weight decreased (Investigations) | 0 (0) | 3 (6) | 5 (6) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 13 (17) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 4 (4)
Dizziness (Nervous system disorders) | 4 (6) | 4 (6) | 5 (6) | 4 (5)
Headache (Nervous system disorders) | 7 (11) | 4 (4) | 10 (13) | 5 (8)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02973100/SAP_000.pdf
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02973100/Prot_001.pdf